CLINICAL TRIAL: NCT06296628
Title: Comparative Study on Mirror Therapy With a Rehabilitation Device for Training of Affected Fingers
Brief Title: Rehabilitation Device for Hand Mirror Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Management Center Innsbruck (MCI), Austria (Unknown); Yale School of Engineering Center for Engineering Innovation and Design (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2000037049; 000 (Other: CTGTY)
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy

STUDY DESIGN:
Intervention Model Description: Participants are patients admitted to the acute inpatient rehabilitation unit for rehabilitation of the hand and fingers who have one paralyzed hand without pronounced spasticity.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Conventional Therapy Group (Active Comparator): Participants in this group with train using Mirror Therapy (MT), the current standard of care.
  Interventions: Behavioral: Mirror Therapy
- Miraπ Group (Experimental): Participants in this group will train with the Miraπ device.
  Interventions: Device: Miraπ

INTERVENTIONS:
Device: Miraπ — This device has tiny sensors that measure the movement of the healthy fingers and tiny motors that move the affected fingers of the patient.
  The device is connected to a specially designed finger mechanism that moves the affected fingers of the patient. This opening mechanism is designed in a way that it prevents the fingers from being forced into any hurting position. If the patient moves the healthy fingers during training, also the fingers of the affected hand are moved by the device at the same time. This creates the effect of mirror therapy for the brain as the patient can see both hands moving.
  Arms: Miraπ Group
Behavioral: Mirror Therapy — Current standard of care using MT.
  Arms: Conventional Therapy Group

SUMMARY:
This study is a randomized and open comparative study that uses two parallel groups: a control group training with conventional therapy and another group that trains with the device "Miraπ". The participants are patients with stroke with motor weakness in one hand. Two measurement visits are required. During those visits, different hand function assessments will be carried out to analyze the motor function of the subjects hand. The measurements will be done during their inpatient rehabilitation stay, one at time of admission and the second at discharge, each taking 20 minutes. In the time between the measurement visits, the hand therapy takes place fivemtimes a week.

DETAILED DESCRIPTION:
The investigators hypothesize that the physical MT with Miraπ with physical movement of the affected hand will be generating a better patient outcome than conventional MT. Until now MT is performed in front of a mirror with the help of an occupational therapist, which can prove to be difficult. The affected hand of the patient is not moved during training. For the reasons mentioned, the mirror therapy device MIRAπ was developed. With MIRAπ, no mirror is needed and the affected hand is also physically moved by the device. Therefore, this clinical trial will focus on evaluating the device to see if it works better than conventional MT and therefore creates greater benefits to the patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants currently accepted and cleared for rehabilitation in the inpatient rehabilitation unit by the rehabilitation medical director.
* Participants with paralysis or motor function problems of only one hand.
* Participants spasticity of the affected hand ( as assessed by by the occupational therapist)
* Participants need mirror therapy because of their health condition.
* Participants are able to memorize easy tasks, and able to follow instructions e.g., moving the healthy fingers.

Exclusion Criteria:

* Participants who are not cleared physically or medically to participate in standard acute inpatient rehabilitation therapies by the rehabilitation medical director
* Participants who are not able to memorize easy tasks, e.g., moving the healthy fingers.
* Participants with spasticity of the affected hand ( as assed by the occupational therapist)
* Vulnerable populations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Change in Jebsen-Taylor Hand Function Test score | At admission and discharge up to 4 weeks
  Percentage score, which determines how well a participant can do motor tasks for range of motion, strength, and tasks of activities of daily life. Participants have up to 120 seconds to complete tasks. Lower scores indicate less impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Rummana Aslam, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Health Inpatient Rehabilitation Unit, Bridgeport Hospital, Bridgeport, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
The plan is to submit abstract of the study to Association of Academic Physiatrists and to publish in peer reviewed engineering and rehabilitation journals. The PI holds the primary responsibility for publishing the study results.